CLINICAL TRIAL: NCT07292116
Title: Prediction of Disease Progression Using Machine Learning Based on Clinical Data in People With Multiple Sclerosis
Brief Title: Disease Progression in ms
Status: Not yet recruiting | Type: Observational
Sponsor: Hüseyin Bektaş (Other)
Responsible Party: Sponsor-Investigator, Hüseyin Bektaş, uzman, Pamukkale University
Organization: Pamukkale University (Other)
Other Study IDs: 53513060613
Record Dates: First submitted 2025-03-12; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Prediction of Disease Progression; Multiple Sclerosis
Keywords: Multiple sclerosis (MS); artificial intelligence; motor learning
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- intervention group

SUMMARY:
Demographic and clinical data will be obtained from people with MS. Based on this data, the progression of the disease will be predicted with artificial intelligence.

DETAILED DESCRIPTION:
Demographic and clinical data will be obtained from people with MS. Demographic data; age, gender, disease type, disease duration. Clinical data; Frailty, Physical Activity Level, Walking, Balance, Fatigue, Quality of Life. Based on these data, disease progression will be predicted with artificial intelligence and motor learning.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with MS

Exclusion Criteria:

* be literate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MS patients coming to Tatvan State Hospital
Sampling Method: Probability Sample
Enrollment: 53 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2025-12-20 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Fragility level | 3 month
  The level of frailty will be measured by the Frailty Index.

IPD SHARING:
Plan to Share IPD: No
The results of the study will be announced